CLINICAL TRIAL: NCT04294121
Title: Testing the Validity of a Novel Method for Identifying and Measuring Child-appealing Marketing on Product Packaging Using Focus Groups of School-aged Children (<13 Years) and Their Parents.
Brief Title: Can a Coding Tool Accurately Evaluate How Kids Respond to Marketing on Food Packaging?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Mary L'Abbe, Professor, University of Toronto
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 37436
Record Dates: First submitted 2020-02-26; First posted 2020-03-03 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Food Marketing
Keywords: food marketing; marketing to children; product packaging; validation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Children (Experimental): Children aged 5-13 years, all genders, will be exposed to a set of breakfast cereals displaying varying child-appealing and parent-appealing marketing techniques as well as varying degrees of child-appealing marketing power on their packaging. Children will be asked to determine if each individual cereal is "child-appealing" (i.e., yes or no). Children will also be asked to rank the cereals in order of their preference (i.e., Most (1) to Least (6)). Children will then participate in a focus group discussion about the why they classified/ranked the cereals the way that they did.
  Interventions: Other: Food marketing on product packaging
- Parents (Experimental): Parents or guardians of the children in the study will be exposed to a set of breakfast cereals displaying varying child-appealing and parent-appealing marketing techniques as well as varying degrees of child-appealing marketing power on their packaging. Parents will be asked to determine if each individual cereal is "child-appealing" (i.e., yes or no). Parents will also be asked to rank the cereals in order of which they would be most likely to purchase for a child (i.e., Most (1) to Least (6)). Parents will then participate in a focus group discussion about the why they classified/ranked the cereals the way that they did.
  Interventions: Other: Food marketing on product packaging

INTERVENTIONS:
Other: Food marketing on product packaging — Participants will be exposed to product packages displaying varying child- and parent-appealing marketing techniques and different degrees of marketing power

SUMMARY:
Child-appealing marketing for unhealthy foods and beverages is a global public health concern, and marketing on product packaging is one of children's top sources of exposure to this type of marketing. However, there is currently no consistent method for evaluating the extent and power of child-appealing marketing on packaging, and therefore, the child-appealing packaging (CAP) coding tool was developed. This study aims to validate this novel tool by testing if the coding tool can accurately evaluate how kids respond to marketing on food packaging. The hypothesis for this study is that the CAP tool will be able to classify and rank marketing on product packaging similarly to how children and their parents rank the same food packages. In order to test this hypothesis, children and their parents will complete an activity where they classify breakfast cereals displaying different degrees of child-appealing marketing power as "child-appealing" or "non-child-appealing" and then rank them in order of their preference. Children and parents will also complete a focus group discussion to talk about why they classified and ranked the cereals the way that they did in the previous activity. Analyses will determine how well participants classifications and rankings agree with the CAP tool's classifications and rankings.

DETAILED DESCRIPTION:
RATIONALE & OBJECTIVES

In Canada, the Child Health Protection Act (Bill S-228) was introduced in September 2016 by Senator Greene Raine to amend the current Food and Drugs Act to prohibit food and beverage marketing directed at children under 13 years of age. Shortly after, to support Bill S-228, Health Canada committed to introducing marketing restrictions as part of its Healthy Eating Strategy. The proposed restrictions will apply to a broad range of marketing platforms, including product packaging, which has been shown to be a top source of children's exposure to food and beverage advertising. Research has also assessed child-appealing marketing within the packaged food environment in Canada; however, these studies are limited due to the significant heterogeneity in the criteria that has been used for identifying child-appealing marketing techniques, with most only recording a few broad techniques, thus hindering their ability to capture the full scope of this marketing practice. Furthermore, despite recommendations from the World Health Organization (WHO) to limit both the exposure and the power of child-appealing marketing, there has been no formal quantification of the power of child-appealing marketing on product packaging.

In response to this gap, the child-appealing packaging (CAP) coding tool was developed to systematically assess the extent, nature and power of child-appealing marketing on product packaging. However, the CAP tool requires formal validation before being implemented in practice. This study will test the criterion and content validity of the CAP tool. Criterion validity is defined as the "extent to which the method is accurately based on an externally derived gold standard; examines whether method correlates in a predicted manner with variables with which, theoretically, it should correlate". Content validity is defined as the "extent to which the system covers the full range of meaning for the concept being measured".

Upon the validation of the CAP tool, its application will enable a comprehensive and updated assessment of the current Canadian marketing environment and be crucial to our ability to continue to accurately track the presence of child-appealing marketing in Canada. Findings from the use of the CAP tool will help inform ongoing policy and regulatory development and provide baseline data from which to monitor the 5-year impact of Bill S-228 as part of the mandatory monitoring period which will be implemented with the legislation.

Objectives: The objectives of this study are to use a product classification activity and focus groups of children and their parents to:

1. Test the criterion validity of the CAP tool by comparing: a) How the CAP tool distinguishes between child-appealing and non-child-appealing products with how children and parents distinguish between these types of products and b) how the CAP tool scores the marketing power of a product's packaging with how children and parents rank their preference of products with child-appealing marketing with varying marketing power
2. Test the content validity of the CAP tool by comparing the marketing techniques included in the tool with the aspects of packaging that children and parents identify as important for appealing to children and parents.

Hypothesis: It is hypothesized that the CAP tool's distinction between child-appealing and non-child-appealing products, scoring of marketing power, and inclusion of marketing techniques will align with how children and parents respond to child-appealing products.

Significance: This research will be conducted as part of a grant funded by the Joannah and Brian Lawson Centre for Child Nutrition entitled "Evaluating Food Environment Policies to Support Healthy Eating among Children" as well as a Project Grant funded by the Canadian Institutes of Health Research entitled "The IMPACT of food environment policies on the Canadian food supply, dietary intakes and health: evidence to inform policy action". The research team will share the results of this study with Health Canada to inform the monitoring of the impact of Bill S-228 on reducing the exposure and power of child-appealing marketing on product packaging. Results will be presented at scientific conferences and published in the peer-reviewed scientific literature. Results will also be shared with the participants through infographics or other lay materials provided to the participating Centres and available on our lab website (labbelab.utoronto.ca).

METHODOLOGICAL OVERVIEW

This mixed methods validation study will compare children and parent's assessments of child-appealing products with the CAP tool's assessments of child-appealing products. This validity testing will be conducted through a brief classification activity, followed by focus group discussions with children and parents. The sessions for children and parents will be conducted separately, but concurrently. Given that the primary goal of the CAP tool is to identify and score marketing on product packaging that may appeal to children, this study will use children to validate the CAP tool's ability to score products that appeal to them. Furthermore, since parents are the primary purchasers of the food that children consume, we aim to validate the CAP tool's ability to score products that may appeal to parents when they are purchasing for their children, as increased marketing to parents may be an unintended consequence of restricting child-appealing marketing.

Child-appealing Packaging (CAP) coding tool: Drawing on a comprehensive list of marketing techniques derived from a review of the scientific literature, the CAP tool was developed to measure the extent, nature and power of child-appealing marketing on product packaging. Despite the knowledge that the number of marketing instances that occur on a package can increase the persuasiveness or intensity of the marketing message, and WHO recommendations to limit both the exposure and power of child-appealing marketing, there has been no formal quantification of marketing power as it relates to child-appealing food and beverage products. The CAP tool provides a novel method for assessing this construct.

Design of sample products: In order to reduce any response bias based on brand-familiarity or preference, a set of 6 mock breakfast cereal packages were designed for use in this study. Cereals were chosen as the example product type given their frequent display of child-appealing marketing on packaging and because they are a food category that is commonly consumed by children. The cereals were designed to portray both child-appealing and non-child appealing marketing with a range of marketing power scores, as would be measured using the CAP tool.

Validation Study Procedures: In order to test the validity of the CAP tool, an independent classification activity will be conducted, followed by separate focus group discussions among children and parents (conducted concurrently).

Children Classification Activity: Children will be welcomed and explained the instructions and expectations all together as a group. Children will then be accompanied one by one to view the set of 6 cereals. A researcher will remind them of the instructions and ask them to decide 1) if each cereal is for children (YES or NO) and 2) to put the cereals in order of which they like the most to which they like the least (1-6). The researcher will record their answers on a response sheet.

Children Focus Group Discussion: Immediately following the completion of the children's classification activity, children will be directed to another room where a focus group discussion will take place. Discussion will prompt children to explain their choices in the classification activity to gain valuable insight into the rationale behind how they classified the cereals in the activity. The moderator will also probe children for examples of aspects of packaging that they think are important for making children like it. A second researcher will record the focus group discussions (audio only) as well as take notes during the discussion to supplement the audio recordings.

Parents Classification Activity: Following the completion of the children's classification activity, parents will be instructed to complete a similar classification activity. A second researcher will facilitate this portion of the study. Parents will be explained the instructions all together as a group and given a response form to fill out. One by one, parents will view the same set of 6 cereals and record 1) if they think each cereal is for children (YES or NO) and 2) their ranking of cereals (1-6) in order of which they would be most likely to purchase for their children to which they would be least likely to purchase for their children.

Parents Focus Group Discussion: Immediately following the completion of the parent's classification activity, parents will be directed to another room where a focus group discussion will take place. Discussion will prompt parents to explain their choices in the classification activity to gain valuable insight into the rationale behind how they classified the cereals in the activity. The moderator will also probe parents for examples of aspects of packaging that they think are important for influencing parents to make purchases for their children. A second researcher will record the focus group discussions (audio only) as well as take notes during the discussion to supplement the audio-recordings.

ELIGIBILITY:
Inclusion Criteria:

* Children: 5-13 years of age
* Parents: must be parents or guardians of children participating in the study
* Must be able to speak/comprehend English
* Must be somewhat familiar with packaged breakfast cereal (e.g., has consumed or seen it before)

Exclusion Criteria:

* N/A

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-05-21 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Kappa agreement between participants' binary ranking of cereals and the child-appealing packaging (CAP) coding tool's binary ranking of cereals | Through study completion, approximately 1 year
  Kappa statistics will evaluate the agreement between how children and parents rank breakfast cereals as either "child-appealing" or "non-child-appealing" and how the CAP tool ranks the same cereals.
Correlation between participants' ordinal ranking of cereals and the child-appealing packaging (CAP) coding tool's ordinal ranking of cereals according to their marketing power. | Through study completion, approximately 1 year
  Spearman Rank Correlation analysis will evaluate the correlation between how children and parents rank breakfast cereals in terms of their ranked preference (children) or ranked purchasing intentions (parents) and how the CAP tool ranks the same cereals according to their marketing power.
Thematic content analysis of focus group transcripts and qualitative agreement with CAP tool | Through study completion, approximately 1 year
  Thematic content analysis will elucidate key themes from the focus group discussions with children and parents, and qualitatively compare them to the contents of the CAP coding tool.

CONTACTS AND LOCATIONS:
Overall Officials: Mary R L'Abbe, PhD, Principal Investigator — University of Toronto
Locations (1):
- University of Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Senate of Canada. Bill S-228: An Act to amend the Food and Drugs Act (prohibiting food and beverage marketing directed at children) - As passed in Senate. First Session, Forty-second Parliament, 64-65-66 Elizabeth II, 2015-2016-2017 ed.; September, 28, 2017. Available from: https://www.parl.ca/DocumentViewer/en/42-1/bill/S-228/third-reading (Accessed Feb 29, 2020)
- [Background] Health Canada. Healthy Eating Strategy. Ottawa, Canada, 2016; p 10. Available from: https://healthycanadians.gc.ca/publications/eating-nutrition/healthy-eating-strategy-canada-strategie-saine-alimentation/alt/pub-eng.pdf (Accessed Feb 29, 2020)
- [Background] Signal LN, Stanley J, Smith M, Barr MB, Chambers TJ, Zhou J, Duane A, Gurrin C, Smeaton AF, McKerchar C, Pearson AL, Hoek J, Jenkin GLS, Ni Mhurchu C. Children's everyday exposure to food marketing: an objective analysis using wearable cameras. Int J Behav Nutr Phys Act. 2017 Oct 8;14(1):137. doi: 10.1186/s12966-017-0570-3. PMID 28988542
- [Background] Elliott, C.D. Packaging fun: Analyzing supermarket food messages targeted at children. Canadian Journal of Communication 2012, 37, 303.
- [Background] Murray, C. Examining the Nutritional Content of Prepackaged Foods and Beverages Marketed to Children in Canada. Unpublished Thesis, University of Toronto, Canada, 2014.
- [Background] Labonte ME, Poon T, Mulligan C, Bernstein JT, Franco-Arellano B, L'Abbe MR. Comparison of global nutrient profiling systems for restricting the commercial marketing of foods and beverages of low nutritional quality to children in Canada. Am J Clin Nutr. 2017 Dec;106(6):1471-1481. doi: 10.3945/ajcn.117.161356. Epub 2017 Oct 25. PMID 29070562
- [Background] World Health Organization. Set of recommendations on the marketing of foods and non-alcoholic beverages to children. 2010; p 16. Available from: https://apps.who.int/iris/bitstream/handle/10665/44416/9789241500210_eng.pdf;jsessionid=0B8A48211C6AA78F83A6482C48838A9C?sequence=1 (Accessed Feb 29, 2020)
- [Background] Townsend MS. Where is the science? What will it take to show that nutrient profiling systems work? Am J Clin Nutr. 2010 Apr;91(4):1109S-1115S. doi: 10.3945/ajcn.2010.28450F. Epub 2010 Feb 17. PMID 20164310
- [Background] Cao, Z.; Yan, R. Health Creates Wealth? The Use of Nutrition Claims and Firm Financial Performance. Journal of Public Policy & Marketing 2016, 35, 58-75, doi:10.1509/jppm.14.142.
- [Background] Mulligan C, Labonte ME, Vergeer L, L'Abbe MR. Assessment of the Canadian Children's Food and Beverage Advertising Initiative's Uniform Nutrition Criteria for Restricting Children's Food and Beverage Marketing in Canada. Nutrients. 2018 Jun 22;10(7):803. doi: 10.3390/nu10070803. PMID 29932134
- [Background] Potvin Kent M, Cameron C, Philippe S. The healthfulness and prominence of sugar in child-targeted breakfast cereals in Canada. Health Promot Chronic Dis Prev Can. 2017 Sep;37(9):266-273. doi: 10.24095/hpcdp.37.9.02. PMID 28902476
- [Background] Subar AF, Krebs-Smith SM, Cook A, Kahle LL. Dietary sources of nutrients among US children, 1989-1991. Pediatrics. 1998 Oct;102(4 Pt 1):913-23. doi: 10.1542/peds.102.4.913. PMID 9755265
- [Background] Fox MK, Condon E, Briefel RR, Reidy KC, Deming DM. Food consumption patterns of young preschoolers: are they starting off on the right path? J Am Diet Assoc. 2010 Dec;110(12 Suppl):S52-9. doi: 10.1016/j.jada.2010.09.002. PMID 21092769
- [Derived] Mulligan C, Potvin Kent M, Vergeer L, Christoforou AK, L'Abbe MR. Quantifying Child-Appeal: The Development and Mixed-Methods Validation of a Methodology for Evaluating Child-Appealing Marketing on Product Packaging. Int J Environ Res Public Health. 2021 Apr 29;18(9):4769. doi: 10.3390/ijerph18094769. PMID 33947116